CLINICAL TRIAL: NCT03481712
Title: Danish Study of Non-Invasive Diagnostic Testing in Coronary Artery Disease 2
Acronym: Dan-NICAD 2
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 000-0001
Record Dates: First submitted 2018-01-25; First posted 2018-03-29 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Angina Pectoris; Atherosclerosis; Coronary Artery Disease; Myocardial Ischemia
MeSH Terms: conditions — Angina Pectoris; Atherosclerosis; Coronary Artery Disease; Myocardial Ischemia | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic tests — Head-to-head comparison between:
  * CADScor and Diamond-Foster score
  * Rb PET and 3T CMRI
  * QFR and ICA-FFR

SUMMARY:
In a cohort of symptomatic patients referred to coronary computed tomography angiography (CCTA), the investigators aim:

1. To investigate and compare the diagnostic precision of Rubidium Positron Emission Tomography (Rb PET) and 3 Tesla Cardiac Magnetic Resonance imaging (3T CMRI) in patients where CCTA does not exclude significant coronary artery disease (CAD) using invasive coronary angiography with fractional flow reserve (ICA-FFR) as reference standard.
2. To evaluate the diagnostic precision of quantitative flow ratio (QFR) and ICA-FFR in patients where CCTA does not exclude significant CAD using Rb PET and 3T CMRI as reference standard.
3. To show superiority for the CADScor®System compared to the Diamond-Forrester score in detection of CAD with CCTA and ICA quantitative coronary angiography (ICA-QCA) as reference standard.
4. To study the diagnostic accuracy of computed tomography fractional flow reserve (CT-FFR) in patients where CCTA does not exclude significant CAD with ICA-FFR as reference standard.
5. To identify and characterize genetic risk variants´ and circulating biomarkers´ importance in developing CAD.
6. To evaluate the bone mineral density in the hip and spine and correlate this to the degree of vascular calcification.

DETAILED DESCRIPTION:
CCTA has become the preferred diagnostic modality for symptomatic patients with low to intermediate risk of CAD. Of the patients examined, CCTA exclude cardiovascular disease in 70-80% with an excellent negative predictive value of more than 95%. Having a low positive predictive value, however, CCTA often overestimates the severity of CAD, especially in patients with moderate to severe coronary calcification. Following CCTA, patients are hence unnecessarily tested using golden standard ICA-FFR. These ICAs often show no obstructive coronary stenosis and are therefore not followed by revascularization. The issues outlined raises the question of whether it is possible (1) to make a more precise risk stratification and consequently better selection of patients prior to CCTA and (2) to reduce the number of patients referred for unnecessary ICAs following CCTA.

In patients with suspicion of coronary stenosis detected by CCTA, current guidelines recommend verification of myocardial ischemia. In Dan-NICAD 2, we intend to investigate the diagnostic accuracy of advanced non-invasive myocardial perfusion imaging tests; Rb PET and 3T CMRI. These examinations have shown a high diagnostic accuracy in symptomatic patients with high risk of ischemic heart disease. However, the diagnostic accuracy is not investigated in patients as follow-up after CCTA.

An alternative way to increase the diagnostic accuracy of CCTA and thus avoid unnecessary downstream testing using ICA is to utilize the ability to extract physiological information from the anatomical CCTA images. CT-FFR has in previous studies shown promising results. CT-FFR has not been head to head compared against Rb PET and 3T CMRI.

Obtained during ICA, QFR is a novel wire-free approach for fast computation of FFR with potential to increase the global use of physiological lesion assessment. QFR is superior to traditional assessment of intermediate coronary lesions (ICA-QCA diameter stenosis). However, disagreement between FFR and QFR has been identified in up to 20% of all measurements.

Acoustic detections of coronary stenosis from automatically recorded and analyzed heart sounds is a newly developed technology potentially useful for pre-test risk stratification before e.g. CCTA. One of these devices, the CADScor®System, has previously shown an area under the receiver operating characteristic curve (AUC of ROC) of 70-80% compared to conventional ICA-QCA. This indicates that the CADScor®System could potentially supplement clinical assessment of CAD and be used for risk stratification prior to CCTA.

The investigators aim to obtain blood samples for biobank purposes and record heart sounds with the CADScor®System in 2000 patients that by clinical evaluation undergo CCTA. In approximately 400 patients (20%), CCTA does not exclude significant CAD. These patients are all examined using Rb PET, 3T CMRI, and ICA with QCA. In patients with a coronary diameter stenosis of 30-90% determined during the ICA examination, FFR, coronary flow reserve (CFR) and QFR is performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for CCTA.
* Qualified patients who have signed a written informed consent form.

Exclusion Criteria:

CADScor specific

* Fragile or compromised skin in the area for application of the CADScor®Patch.
* Known allergy to polyacrylate adhesives.
* Significant operation scars or abnormal body shape in left IC4 (4th Inter Costal region).
* Use of vasodilating agents at the same day and prior to CAD-score measurements.

Demography and co-existing cardiac morbidity specific

* Age below 30 years.
* Patients having a donor heart, a mechanic heart, or mechanical heart pump.
* Suspicion acute coronary syndrome Previous revascularization.

Scan specific

CCTA:

* Pregnant women, including women who are potentially pregnant or lactating.
* Reduced kidney function, with an estimated glomerular filtration rate (eGFR) < 40 mL/min.
* Allergy to X-ray contrast medium.

CMRI and PET:

* Contra-indication for adenosine (severe asthma, advanced AV block, or critical aorta stenosis).
* Contra-indications for MRI (implanted medicinal pumps or nerve stimulators, magnetic foreign objects in sensitive areas, i.e. the eye).
* Patients having an ICD or pacemaker, a cochlea implant, or metal clips evaluated by the including doctor.

General:

- Patients not able to breath-hold (COPD/asthma).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for CCTA.
Sampling Method: Probability Sample
Enrollment: 1732 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of 3T CMRI vs. Rb PET. | 4 weeks after inclusion.
  Head-to-head comparison using ICA-FFR as reference standard. Diagnostic accuracy is measured using specificity, sensitivity, positive and negative predictive value and likelihood ratios.
Diagnostic accuracy of QFR vs. ICA-FFR. | 4 weeks after inclusion.
  Head-to-head comparison using myocardial perfusion examinations as reference standard.
  Diagnostic accuracy is measured using specificity, sensitivity, positive and negative predictive values, likelihood ratios and area under receiving operating curves (AUC-ROC).
Diagnostic accuracy of CADScor vs. Diamond-Foster Score. | 4 weeks after inclusion.
  AUC-ROC for CAD-score and Diamond-Forrester score in detection of CAD with CCTA and ICA-QCA as reference in patients ≥40 years.

SECONDARY OUTCOMES:
Genome-wide Associations. | 4 weeks after inclusion.
  The primary analysis will be a genome-wide association analysis, to determine candidate genes and markers underlying coronary artery disease and bone mineralization.
Bone mineral density. | 1 day after inclusion.
  To study the bone mineral density in this cohort and its relation to vascular calcification.
Coronary flow measurement´s impact on diagnostic accuracy of myocardial perfusion imaging (MPI). | 4 weeks after inclusion.
  Impact of coronary flow reserve (CFR) and index of microcirculatory resistance (IMR) on myocardial perfusion imaging (MPI) diagnostic accuracy using specificity, sensitivity, positive and negative predictive values.
Diagnostic accuracy of quantitative CMRI analysis. | 4 weeks after inclusion.
  Diagnostic accuracy of quantitative CMRI analysis compared to ICA with FFR-CFR.
Absolute measurements of coronary flow with quantitative CMRI analysis. | 4 weeks after inclusion.
  Correlation analysis between flow measurements estimated by quantitative CMRI vs. Rb PET.
Diagnostic accuracy of CADScor vs. Diamond-Foster Score. | 4 weeks after inclusion.
  AUC-ROCs for CAD-score and Diamond-Forrester score in detection of CAD with CCTA and ICA-QCA as reference in total population.
Diagnostic accuracy of CADScor vs. Diamond-Forrester Score. | 4 weeks after inclusion.
  Sensitivity, specificity, negative and positive predictive value of CAD-score and Diamond-Forrester score with CCTA and ICA-QCA as reference standard.
  For the CADScor®System specifically, the following criteria are applicable:
  * Sensitivity >79%
  * Negative predictive value maximum 3% lower than the anticipated negative predictive value
  * Rule-out proportion ≥30%
CADScor. | 4 weeks after inclusion.
  AUC-ROCs, sensitivity, specificity, negative and positive predictive value of CAD-score with ICA-FFR as reference standard.
QFR FFR mismatch. | 4 weeks after inclusion.
  A subgroup analysis is performed for patients with mismatch between QFR and FFR using CFR and IMR as reference standard.
Diagnostic accuracy of CT-FFR. | 4 weeks after inclusion.
  To evaluate the diagnostic accuracy of CT-FFR using ICA-FFR as reference standard.
Effect of revascularisation on symptoms of angina pectoris. | 3+12 months after ICA
  Evaluation of coronary revascularissation to reduce symptoms of angina pectoris 3 and 12 mdr. after ICA.
Prognostic value of clinical, biomarker, and genetic information. | 3+5+10 years after inclusion.
  To validate the 3, 5 and 10 yr. prognostic value of a pre-test probability score including clinical, biomarker and genitic information in patients with symptoms suggestive of CAD referred for coronary CTA.
Prognostic value of heart sound analysis and CAD-score. | 3+5+10 years after inclusion.
  To investigate the 3, 5 and 10 yr. prognostic value of pre-specified heart sound analysis and CAD-score in patients with symptoms suggestive of CAD referred for coronary CTA.
Prognostic value of coronary CTA, RbPET, 3T CMR, CT-FFR and QFR | 3+5+10 years after inclusion.
  To investigate the 3, 5 and 10 yr. prognostic value of the study's imaging techniques in patients with symptoms suggestive of CAD referred for coronary CTA.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Böttcher, MD, Ph.D, Principal Investigator — Regional Hospital of Herning, department of cardiology
Locations (5):
- Denmark (5):
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Regional Hospital of Herning, Herning, Central Jutland
  - Regional Hospital of Silkeborg, Silkeborg, Central Jutland
  - Regional Hospital of Randers, Randers
  - Regional Hospital of Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rasmussen LD, Sikjaer M, Soby JH, Pedersen OB, Westra J, Efthekhari A, Christiansen EH, Foldyna B, Williams MC, Dweck MR, Newby DE, Douglas PS, Bottcher M, Winther S. Dual probability approach for risk adjustment in patients with a low clinical likelihood of coronary artery disease. Eur Heart J Cardiovasc Imaging. 2025 Aug 29;26(9):1507-1517. doi: 10.1093/ehjci/jeaf193. PMID 40590244
- [Derived] Brix GS, Rasmussen LD, Rohde PD, Nissen L, Nyegaard M, O'Donoghue ML, Bottcher M, Winther S. Elevated lipoprotein(a) levels are independently associated with the presence of significant coronary stenosis in de-novo patients with stable chest pain. Am Heart J. 2025 Apr;282:103-113. doi: 10.1016/j.ahj.2025.01.001. Epub 2025 Jan 7. PMID 39788470
- [Derived] Karim SR, Westra JS, Rasmussen LD, Eftekhari A, Sejr-Hansen M, Winther S, Bottcher M, Christiansen EH. Effect of Guiding Catheter Extubation During Physiological Assesment of Stenosis. Catheter Cardiovasc Interv. 2025 Mar;105(4):735-744. doi: 10.1002/ccd.31370. Epub 2024 Dec 30. PMID 39736151
- [Derived] Rasmussen LD, Westra J, Karim SR, Dahl JN, Soby JH, Ejlersen JA, Gormsen LC, Eftekhari A, Christiansen EH, Bottcher M, Winther S. Microvascular resistance reserve: impact on health status and myocardial perfusion after revascularization in chronic coronary syndrome. Eur Heart J. 2025 Feb 3;46(5):424-435. doi: 10.1093/eurheartj/ehae604. PMID 39217607
- [Derived] Rasmussen LD, Murphy T, Milidonis X, Eftekhari A, Karim SR, Westra J, Dahl JN, Isaksen C, Brix L, Ejlersen JA, Nyegaard M, Johansen JK, Sondergaard HM, Mortensen J, Gormsen LC, Christiansen EH, Chiribiri A, Petersen SE, Bottcher M, Winther S. Myocardial Blood Flow by Magnetic Resonance in Patients With Suspected Coronary Stenosis: Comparison to PET and Invasive Physiology. Circ Cardiovasc Imaging. 2024 Jun;17(6):e016635. doi: 10.1161/CIRCIMAGING.124.016635. Epub 2024 Jun 18. PMID 38889213
- [Derived] Rasmussen LD, Gormsen LC, Ejlersen JA, Karim SR, Westra J, Knudsen LL, Kirk J, Sondergaard HM, Mortensen J, Knuuti J, Christiansen EH, Eftekhari A, Bottcher M, Winther S. Impact of Absolute Myocardial Blood Flow Quantification on the Diagnostic Performance of PET-Based Perfusion Scans Using 82Rubidium. Circ Cardiovasc Imaging. 2024 Jan;17(1):e016138. doi: 10.1161/CIRCIMAGING.123.016138. Epub 2024 Jan 16. PMID 38227687
- [Derived] Rasmussen LD, Winther S, Eftekhari A, Karim SR, Westra J, Isaksen C, Brix L, Ejlersen JA, Murphy T, Milidonis X, Nyegaard M, Benovoy M, Johansen JK, Sondergaard HM, Hammid O, Mortensen J, Knudsen LL, Gormsen LC, Christiansen EH, Chiribiri A, Petersen SE, Bottcher M. Second-Line Myocardial Perfusion Imaging to Detect Obstructive Stenosis: Head-to-Head Comparison of CMR and PET. JACC Cardiovasc Imaging. 2023 May;16(5):642-655. doi: 10.1016/j.jcmg.2022.11.015. Epub 2023 Feb 8. PMID 36881421
- [Derived] Rasmussen LD, Winther S, Karim SR, Westra J, Kirk Johansen J, Sondergaard HM, Hammid O, Sevestre E, Onuma Y, Nyegaard M, Ejlersen JA, Hoj Christiansen E, Eftekhari A, Holm NR, Schmidt SE, Bottcher M. Likelihood reclassification by an acoustic-based score in suspected coronary artery disease. Heart. 2023 Jul 27;109(16):1223-1230. doi: 10.1136/heartjnl-2023-322357. PMID 36878672
- [Derived] Rasmussen LD, Winther S, Westra J, Isaksen C, Ejlersen JA, Brix L, Kirk J, Urbonaviciene G, Sondergaard HM, Hammid O, Schmidt SE, Knudsen LL, Madsen LH, Frost L, Petersen SE, Gormsen LC, Christiansen EH, Eftekhari A, Holm NR, Nyegaard M, Chiribiri A, Botker HE, Bottcher M. Danish study of Non-Invasive testing in Coronary Artery Disease 2 (Dan-NICAD 2): Study design for a controlled study of diagnostic accuracy. Am Heart J. 2019 Sep;215:114-128. doi: 10.1016/j.ahj.2019.03.016. Epub 2019 May 1. PMID 31323454